CLINICAL TRIAL: NCT02323828
Title: Effect of High Resistant Starch-cookies on Food Ingestion and Appetite Control in a Cohort of Healthy Students
Brief Title: High Resistant Starch (RS) Cookies and Appetite Control
Acronym: RS
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Catholic University of the Sacred Heart (Other)
Responsible Party: Principal Investigator, Filippo Rossi, researcher, Catholic University of the Sacred Heart
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 24238/14
Record Dates: First submitted 2014-12-15; First posted 2014-12-24 (Estimated); Last update posted 2016-01-27 (Estimated); Status verified 2016-01

CONDITIONS: Metabolic Syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Investigational product (Experimental): The investigational products are RS starch cookies (40 g resistant starch) from high amylose maize starch.
  Nine young healthy volunteers (males and females) consumed RS rich cookies (40 g RS) in two separate occasions.
  Interventions: Dietary Supplement: High RS cookies
- Placebo (Placebo Comparator): The placebo products are common wheat-maize cookies (2 g RS). Nine young healthy volunteers (males and females) consumed placebo in two separate occasions.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: High RS cookies — High RS cookies ingestion in healthy young adults
  Arms: Investigational product
Dietary Supplement: Placebo — Placebo cookies ingestion in healthy young adults
  Arms: Placebo

SUMMARY:
Evaluation of the effect of ingestion of high RS-cookies prepared from high amylose corn starch on food intake and appetite control of a cohort of healthy students. Cookies were prepared with increasing RS content and were fed to 18 healthy students in a blind trial versus a placebo.

Parameters of interest were: short and long time intake (ad libitum test meal and 12 h diet diaries, respectively).

ELIGIBILITY:
Inclusion Criteria:

* self-reported healthy
* not suffering disorders of lipid metabolism and eating disorders

Exclusion Criteria:

* pregnant or breast-feeding
* consuming an energy-restricted diet
* vegan or vegetarians

Ages: 20 Years to 24 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2013-01; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Consumption of RS on appetite regulation | One day
  Ad libitum test meal
Consumption of RS on appetite regulation | One day
  12-h diet diaries